CLINICAL TRIAL: NCT06179277
Title: Effect of Enamel Matrix Derivative (Emdogain®) on Soft Tissue Wound Healing Following Surgical Crown Lengthening Procedures
Brief Title: Effect of Emdogain® on Soft Tissue Wound Healing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amir Azarpazhooh (Other)
Collaborators: Institut Straumann AG (Industry)
Responsible Party: Sponsor-Investigator, Amir Azarpazhooh, Professor, University of Toronto
Organization: University of Toronto (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 37028
Record Dates: First submitted 2023-12-11; First posted 2023-12-21 (Actual); Last update posted 2023-12-21 (Actual); Status verified 2023-12

CONDITIONS: Periodontal Inflammation; Crown Lengthening

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: All participants remained blinded with respect to their group assignment for the duration of the study. Allocation concealment was done by placing randomization codes with group assignment in opaque sealed envelopes that were opened by the operator at the end of the surgical procedure, right before suturing, which means the surgeon was blinded throughout most of the treatment.
  Data was collected by a separate examiner who was also blinded to treatment allocation. Data analysis was carried out by an external statistician, minimizing the risk of bias.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment/experimental group (Experimental): Patients undergoing surgical crown lengthening of a single site with application of PrefGel® + Emdogain®
  Interventions: Device: PrefGel® + Emdogain®
- Control group (Placebo Comparator): Patients undergoing surgical crown lengthening of a single site with application of PrefGel® only
  Interventions: Device: PrefGel®

INTERVENTIONS:
Device: PrefGel® + Emdogain® — Surgical crown lengthening procedure with root conditioning with 24% EDTA (PrefGel®) and application of 0.3 mL Emdogain® to root surface with 27-gauge needle
  Arms: Treatment/experimental group
Device: PrefGel® — Surgical crown lengthening procedure with root conditioning with 24% EDTA (PrefGel®)
  Arms: Control group

SUMMARY:
The goal of this randomized, controlled, single-center study is to compare the effects of Emdogain®, a regenerative biomaterial, on post-operative pain, wound healing and inflammation of treated sites after surgical crown lengthening. The main question it aims to answer is:

Does the use of Emdogain® in conjunction with crown lengthening surgery improve post-operative soft-tissue healing, decrease inflammation and reduce patient perception of pain compared to crown lengthening without addition of Emdogain®? The treatment group will receive Emdogain® during surgery, and the control group will undergo standard crown lengthening without Emdogain®.

DETAILED DESCRIPTION:
This randomized, controlled, single-center study intends to investigate the effects of Emdogain® on wound healing, postoperative pain and inflammation of treated sites after crown lengthening procedures on a single site, and to compare the results of this therapy with those of standard crown lengthening treatment on a single site. We have hypothesized that the use of Emdogain® in conjunction with crown lengthening surgery improves post-operative soft-tissue healing, decreases inflammation and reduces patient perception of pain compared to crown lengthening without addition of Emdogain®. Patients were recruited from the Graduate Periodontology clinic at the Faculty of Dentistry, University of Toronto. These patients were referred to the department by dental students in the faculty as well as dentists and dental specialists within the community for crown lengthening surgery, and were subsequently screened for eligibility to participate in the study. After confirmation of eligibility and completion of recruitment, patients were randomized, using a computer-generated randomization table, into the following groups:

* Treatment/experimental group: patients undergoing surgical crown lengthening of a single site with application of PrefGel® + Emdogain®
* Control group: patients undergoing surgical crown lengthening of a single site with application of PrefGel® only

ELIGIBILITY:
Inclusion Criteria:

Patients who:

* Were capable and willing to provide consent and complete treatment as well as follow-up appointments
* Were over the age of 18 years old
* Required surgical crown lengthening for functional reasons as outlined in background
* Had no contraindications to surgery (these include periodontal contraindications to crown lengthening such as poor crown-to-root ratio, furcation exposure or esthetic concerns)

Exclusion Criteria:

* Patients who were unable to provide informed consent
* Pregnant women
* Women receiving estrogen therapy
* Patients who had received systemic antibiotics within the past 6 months
* Patients with severe systemic disease (ASA 3+) including: poorly controlled diabetes, blood dyscrasias, liver disease, immunosuppressive disorders, malignancy or who have had previous radiotherapy
* Patients with untreated, active periodontal disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2019-04-08 (Actual); Primary Completion 2020-11-09 (Actual); Study Completion 2021-10-11 (Actual)

PRIMARY OUTCOMES:
Clinician-reported degree of inflammation | One, two, four and eight-week follow-ups
  Presence and degree of inflammation (appearance of erythema/edema) using VAS score
Clinician-reported quality of healing | One, two, four and eight-week follow-ups
  Overall healing using VAS score
Patient-reported perception of pain | One, two, four and eight-week follow-ups
  Pain score using VAS
Patient-reported swelling | One, two, four and eight-week follow-ups
  Swelling score using VAS

SECONDARY OUTCOMES:
Number of analgesics | One, two, four and eight-week follow-ups
  Number of analgesics taken by each participant post-operatively

CONTACTS AND LOCATIONS:
Overall Officials: Howard Tenenbaum, Dr, Principal Investigator — University of Toronto
Locations (1):
- University of Toronto, Faculty of Dentistry, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No